CLINICAL TRIAL: NCT04127786
Title: Immunogenicity and Safety of a Purified Vero Rabies Vaccine - Serum Free in Comparison With Verorab® and Imovax® Rabies, in a Pre-exposure Regimen in Both Pediatric and Adult Populations and a Single Booster Dose of Purified Vero Rabies Vaccine - Serum Free Administered at 1 Year Post-3-dose Primary Series, and Between 2 up to 3 Years Post-One Week 2-Dose Primary Series in a Subset of Adults in Thailand
Brief Title: Study of Purified Vero Rabies Vaccine Compared With Two Reference Rabies Vaccines, Given in a Pre-exposure Regimen to Children and Adults and as Single Booster Dose to a Subset of Adults
Acronym: VRV12
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VRV12; U1111-1217-3241 (Registry Identifier: ICTRP); VRV12 (Other: Sanofi Identifier); 2019-000973-22 (EudraCT Number)
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Rabies; Healthy Volunteers
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Intervention Model Description: Primary series will be observer-blinded for both Cohort 1 (3-dose pre-exposure prophylaxis [PrEP] regimen) and Cohort 2 (one week 2-dose PrEP regimen).
  Booster phase will be conducted in a blinded manner (vaccine received in the primary series) with an adult subset from Cohort 1 and hereafter referred as "Booster Phase Cohort 1" (with booster dose 1 year after the 1st primary series vaccine injection).
  Evaluation of immunogenicity persistence after primary series and a booster phase will be conducted in an open label manner with an adult subset from Cohort 2 and hereafter referred as "Immunogenicity Persistence and Booster Phase Cohort 2" (including blood samples collection at Month 6, Month 12, Month 18, pre-booster between Month 24 up to Month 36, and post-booster between Month 24 up to Month 36+Day 14; and a booster dose between Month 24 up to Month 36).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For cohort 1 primary series and booster dose and cohort 2 primary series. The study is conducted in an observer-blind manner. Unblinded staff members, independent of the safety evaluation and other study evaluations, prepare and administer the vaccine. The Investigator or delegate in charge of safety assessment as well as the participants are blinded and do not know which vaccine is administered.
  In addition to the participants, health care providers, data collectors, outcome assessors (eg, Investigator who assess the safety), the Sponsor personnel (eg, Clinician, Data Management, Biostatistician) will remain blinded until the first statistical analysis.
  For cohort 2 immunogenicity persistence and booster phase This phase is open label, however, the laboratory analysts who will be involved in the blood sample testing will remain blinded during the whole study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group1:VRVg2 Cohort1(C1)-1ry Series:pediatric&adult participants-Booster:102 adult participants (Experimental): VRVg-2, 3 injections at Day 0, Day 7, and Day 28
  Booster dose of VRVg-2 for a subset of 102 adult participants at Month 12
  Interventions: Biological: Purified vero rabies vaccine - serum free - VRVg-2
- Group 2:Verorab C1-1ry Series:pediatric&adult participants-Booster Phase:34 adult participants (Active Comparator): Verorab, 3 injections at Day 0, Day 7, and Day 28
  Booster dose of VRVg-2 for a subset of 34 adult participants at Month 12
  Interventions: Biological: Purified vero rabies vaccine - serum free - VRVg-2; Biological: Purified inactivated rabies vaccine - Verorab®
- Group 3:Imovax Rabies C1-1ry Series:pediatric&adult participants-Booster Phase:34 adult participants (Active Comparator): Imovax Rabies, 3 injections at Day 0, Day 7, and Day 28
  Booster dose of VRVg-2 for a subset of 34 adult participants at Month 12
  Interventions: Biological: Purified vero rabies vaccine - serum free - VRVg-2; Biological: Purified inactivated rabies vaccine - Imovax® Rabies
- Group 4:VRVg-2 Cohort 2(C2)-1ry Series:Adult participants-Booster Phase:138 adult participants (Experimental): VRVg-2, 2 injections at Day 0 and Day 7
  Booster dose of VRVg-2 for a subset of 138 adult participants between Month 24 up to Month 36
  Interventions: Biological: Purified vero rabies vaccine - serum free - VRVg-2
- Group 5:Verorab C2-1ry Series:adult participants-Booster Phase:46 adult participants (Active Comparator): Verorab, 2 injections at Day 0 and Day 7
  Booster dose of VRVg-2 for a subset of 46 adult participants between Month 24 up to Month 36
  Interventions: Biological: Purified vero rabies vaccine - serum free - VRVg-2; Biological: Purified inactivated rabies vaccine - Verorab®
- Group 6:Imovax Rabies C2-1ry Series:adult participants-Booster Phase:46 adult participants (Active Comparator): Imovax Rabies, 2 injections at Day 0 and Day 7
  Booster dose of VRVg-2 for a subset of 46 adult participants between Month 24 up to Month 36
  Interventions: Biological: Purified vero rabies vaccine - serum free - VRVg-2; Biological: Purified inactivated rabies vaccine - Imovax® Rabies

INTERVENTIONS:
Biological: Purified vero rabies vaccine - serum free - VRVg-2 — Pharmaceutical form: Freeze-dried Route of administration: Intramuscular
Biological: Purified inactivated rabies vaccine - Verorab® — Pharmaceutical form:Freeze-dried Route of administration: Intramuscular
  Arms: Group 2:Verorab C1-1ry Series:pediatric&adult participants-Booster Phase:34 adult participants; Group 5:Verorab C2-1ry Series:adult participants-Booster Phase:46 adult participants
Biological: Purified inactivated rabies vaccine - Imovax® Rabies — Pharmaceutical form: Freeze-dried Route of administration: Intramuscular
  Arms: Group 3:Imovax Rabies C1-1ry Series:pediatric&adult participants-Booster Phase:34 adult participants; Group 6:Imovax Rabies C2-1ry Series:adult participants-Booster Phase:46 adult participants

SUMMARY:
The primary objective of this study is:

To demonstrate the VRVg-2 is non-inferior to Verorab and Imovax Rabies vaccines in each age group (pediatric and adult populations) when administered as a 3-dose PrEP regimen, in terms of proportion of participants achieving a rabies virus neutralizing antibody (RVNA) titer ≥ 0.5 IU/mL at Day 42, ie. 14 days after the 3rd injection (for Primary Series Cohort 1).

The secondary objectives of this study are: First 1-5 with hypotheses testing will be evaluated sequentially - only if the previous objective is achieved, will the next objective be tested

To demonstrate that:

* the observed proportion of participants in the VRVg2(VRVg) group at D42 is at least 99% with a lower limit of the 95% confidence interval (CI) of at least 97%
* VRVg is non inferior (NI) to Verorab and Imovax Rabies vaccines (Imovax) in each age group at D28
* 2-dose VRVg at D28 is NI to 3-dose Imovax at D42 in each age group
* the observed proportion of participants in the VRVg group at D28 is at least 99% with a lower limit of the 95% CI of at least 97%
* 2-dose Imovax at D28 is NI to 3-dose Imovax at D42 in overall participants (Cohort1)

To describe:

* the immune response induced by VRVg versus Verorab and Imovax at D28 and at D42 in all age groups
* the immune response induced by VRVg at D14 after a booster dose of VRVg administered at M12 (Cohort1) and between M24 up to M36 (Cohort2)
* the persistence of immune response at M6,12,18, and pre-booster between M24 up to M36 post-primary series vaccination (Cohort2)
* safety profile of VRVg versus Verorab and Imovax in primary series and after a booster dose of VRVg

DETAILED DESCRIPTION:
The duration of each participant's participation in the primary series Cohort 1 of the study will be approximately 7 months (28 day-vaccination period followed by 6-month safety follow-up period). For the subset of adult participants in Booster Phase Cohort 1 who received a single booster dose of VRVg-2 (1 booster dose 365 days after primary series followed by 6-month safety follow-up period), the duration will be approximately 18 months.

For Primary Series Cohort 2, the duration of each participant's participation in the study will be approximately 7 months (one week vaccination period followed by 6-month safety follow-up period).

For the subset of adult participants in Immunogenicity Persistence and Booster Phase Cohort 2 who will be followed-up for evaluation of immunogenicity persistence after primary series (including blood samples collection at M6, M12, M18, and between 24 up to 36 months) and who will receive a single booster dose of VRVg-2 (after the blood sample collection between 24 up to 36 months), the duration will be approximately 30 to 42 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥1 year on the day of inclusion

  * Cohort 1 - pediatrics (>1 to 17 years old) and adult (≥18 years old)
  * Cohort 2 - all adults (≥18 years old)
* Informed consent form has been signed and dated by the participant and /or and parent(s) or legally acceptable representative (LAR) and by an independent witness (if required by local regulations), as necessary; and assent form has been signed and dated by the participant, as required
* Participant (adult ≥18 years) or participant and parent/LAR (1 year to <18 years) are able to attend all scheduled visits and to comply with all study procedures.

Exclusion Criteria:

* Participant is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until 1 month after each vaccination. To be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, or surgically sterile.
* Participation at the time of study enrollment or, planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the first study vaccination or planned receipt of any vaccine prior to Visit 5 for pediatric participants and adult participants in Cohort 1, and prior to Visit 4 for adult participants in Cohort 2.
* Previous vaccination against rabies (in pre- or post-exposure regimen) with either the study vaccines or another vaccine.
* Bite by, or exposure to a potentially rabid animal in the previous 6 months with or without post-exposure prophylaxis.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* At high risk for rabies exposure during the study.
* Known systemic hypersensitivity to any of the study/control vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances.
* Self-reported thrombocytopenia, contraindicating intramuscular vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol or substance abuse that, in the opinion of the investigator, might interfere with the study conduct or completion.
* Chronic illness(1) that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Personal history of Guillain-Barré syndrome.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

  1. Chronic illness may include, but is not limited to, neurological, cardiopulmonary, gastrointestinal, renal, genitourinary, metabolic, hematologic, auto-immune, or psychiatric disorders or infection

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1708 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2025-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (4):
- Thailand (4):
  - Investigational Site Number : 7640001, Bangkok
  - Investigational Site Number : 7640004, Bangkok
  - Investigational Site Number : 7640003, Bangkok
  - Investigational Site Number : 7640002, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Chokephaibulkit K, Huoi C, Tantawichien T, Mootsikapun P, Kosalaraksa P, Kiertiburanakul S, Ratanasuwan W, Vangelisti M, Laot T, Huang Y, Petit C, Pineda-Pena AC, Frago C. Noninferiority Study of Purified Vero Rabies Vaccine-Serum Free in 3-dose and 2-dose Preexposure Prophylaxis Regimens in Comparison With Licensed Rabies Vaccines. Clin Infect Dis. 2025 Oct 6;81(3):654-666. doi: 10.1093/cid/ciae581. PMID 39587931
- See also: VRV12 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25383&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants at 4 active sites in Thailand from 21 October 2019 to 23 January 2023. A total of 1708 participants were enrolled and randomized in the study. The study involves 2 phases: Primary series (Cohort 1: 3-dose pre-exposure prophylaxis [PrEP] regimen and Cohort 2: 1-week 2-dose PrEP regimen); and Booster Phase (Cohort 1: booster dose 1 year after first primary series vaccine injection and Cohort 2: Immunogenicity Persistence and Booster Phase Cohort 2).
Pre-assignment Details: The analysis contains all data in the primary series and booster phase of Cohort (C)-1 and Cohort-2.
Groups:
- Cohort-1 Group 1: VRVg-2/VRVg-2: Pediatric and adult participants received 3 intramuscular (IM) injections of Purified Vero Rabies Vaccine - Serum Free (VRVg-2) vaccine at Day 0, Day 7, and Day 28 respectively in the primary series. A subset of adult participants who received VRVg-2 vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase at Month 12.
- Cohort-1 Group 2: Verorab®/VRVg-2: Pediatric and adult participants received 3 IM injections of Verorab® vaccine at Day 0, Day 7, and Day 28 respectively in the primary series. A subset of adult participants who received Verorab® vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase at Month 12.
- Cohort-1 Group 3: Imovax Rabies®/VRVg-2: Pediatric and adult participants received 3 IM injections of Imovax Rabies® vaccine at Day 0, Day 7, and Day 28 respectively in primary series. A subset of adult participants who received Imovax Rabies® vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase at Month 12.
- Cohort-2 Group 4: VRVg-2/VRVg-2: Adult participants received 2 IM injections of VRVg-2 vaccine at Day 0, and Day 7 respectively in the primary series. A subset of adult participants who received VRVg-2 vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase between Month 24 up to Month 36.
- Cohort-2 Group 5: Verorab®/VRVg-2: Adult participants received 2 IM injections of Verorab® vaccine at Day 0, and Day 7 respectively in the primary series. A subset of adult participants who received Verorab® vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase between Month 24 up to Month 36.
- Cohort-2 Group 6: Imovax Rabies®/VRVg-2: Adult participants received 2 IM injections of Imovax Rabies® vaccine at Day 0, and Day 7 respectively in the primary series. A subset of adult participants who received Imovax Rabies® vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase between Month 24 up to Month 36.
Period: Primary: C-1: Day[D]0-D28; C-2:D0-D7
Arm/Group | Cohort-1 Group 1: VRVg-2/VRVg-2 | Cohort-1 Group 2: Verorab®/VRVg-2 | Cohort-1 Group 3: Imovax Rabies®/VRVg-2 | Cohort-2 Group 4: VRVg-2/VRVg-2 | Cohort-2 Group 5: Verorab®/VRVg-2 | Cohort-2 Group 6: Imovax Rabies®/VRVg-2
Started | 607 | 203 | 200 | 420 | 139 | 139
Safety Analysis Set (SafAS) (SafAS included participant who had received at least one dose of the study vaccine and were analyzed according to the actual treatment received.) | 607 | 202 | 200 | 419 | 139 | 139
Per-protocol Analysis Set (PPAS) for Day 28 (PPAS for Day 28 included all participants who received at least 1 dose of the study vaccine in the primary series, with no relevant protocol deviation before Day 28.) | 519 | 169 | 160 | 342 | 120 | 124
Completed (Completed the active phase of Primary series.) | 599 | 199 | 196 | 415 | 137 | 138
Not Completed | 8 | 4 | 4 | 5 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 5 | 3 | 4 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 2 | 1 | 0 | 0 | 0 | 0
Period: Booster:C-1:At Month(M) 12; C-2:M24-M36
Arm/Group | Cohort-1 Group 1: VRVg-2/VRVg-2 | Cohort-1 Group 2: Verorab®/VRVg-2 | Cohort-1 Group 3: Imovax Rabies®/VRVg-2 | Cohort-2 Group 4: VRVg-2/VRVg-2 | Cohort-2 Group 5: Verorab®/VRVg-2 | Cohort-2 Group 6: Imovax Rabies®/VRVg-2
Started | 94 (Adult participants who completed the follow-up period, entered the booster phase and received booster dose of VRVg-2.) | 31 (Adult participants who completed the follow-up period, entered the booster phase and received booster dose of VRVg-2.) | 32 (Adult participants who completed the follow-up period, entered the booster phase and received booster dose of VRVg-2.) | 128 (Adult participants who completed the follow-up period, entered the booster phase and received booster dose of VRVg-2.) | 41 (Adult participants who completed the follow-up period, entered the booster phase and received booster dose of VRVg-2.) | 43 (Adult participants who completed the follow-up period, entered the booster phase and received booster dose of VRVg-2.)
SafAS | 94 | 31 | 32 | 128 | 41 | 43
Completed | 92 | 31 | 32 | 127 | 41 | 43
Not Completed | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants in the primary series cohorts.
Groups:
- Primary Series: Cohort-1 Group 1: VRVg-2: Pediatric and adult participants received 3 IM injections of VRVg-2 vaccine at Day 0, Day 7, and Day 28 respectively.
- Primary Series: Cohort-1 Group 2: Verorab®: Pediatric and adult participants received 3 IM injections of Verorab® vaccine at Day 0, Day 7, and Day 28 respectively.
- Primary Series: Cohort-1 Group 3: Imovax Rabies®: Pediatric and adult participants received 3 IM injections of Imovax Rabies® vaccine at Day 0, Day 7, and Day 28 respectively.
- Primary Series: Cohort-2 Group 4: VRVg-2: Adult participants received 2 IM injections of VRVg-2 vaccine at Day 0, and Day 7 respectively.
- Primary Series: Cohort-2 Group 5: Verorab®: Adult participants received 2 IM injections of Verorab® vaccine at Day 0, and Day 7 respectively.
- Primary Series: Cohort-2 Group 6: Imovax Rabies®: Adult participants received 2 IM injections of Imovax Rabies® vaccine at Day 0, and Day 7 respectively.
- Total: Total of all reporting groups
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies® | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies® | Total
Number analyzed (Participants) | 607 | 203 | 200 | 420 | 139 | 139 | 1708
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.9 (17.1) | 22.6 (16.1) | 22.4 (16.1) | 37.4 (11.3) | 38.4 (11.1) | 37.3 (10.9) | 28.8 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 399 | 147 | 122 | 266 | 96 | 98 | 1128
  Male | 208 | 56 | 78 | 154 | 43 | 41 | 580
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 607 | 203 | 200 | 420 | 139 | 139 | 1708
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Primary Series Cohort 1: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.5 IU/mL
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method.
Time Frame: Cohort 1: Day 0 (pre-vaccination), Day 28 and Day 42 (post-vaccination)
Population: Analysis was performed on the PPAS for Day 42. Here, 'number analyzed' signifies participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies®
Number analyzed (Participants) | 519 | 169 | 162
percentage of participants
  Day 0 | 0 [0 to 0.7] | 0 [0 to 2.2] | 0 [0 to 2.3]
  Day 28: number analyzed (Participants) | 512 | 168 | 160
  Day 28 | 100 [99.3 to 100] | 99.4 [96.7 to 100] | 98.8 [95.6 to 99.8]
  Day 42 | 100 [99.3 to 100] | 99.4 [96.7 to 100] | 100 [97.7 to 100]
Statistical Analysis 1: Comparison: Primary Series: Cohort-1 Group 1: VRVg-2; The secondary immunogenicity outcome measures were evaluated sequentially following a fixed-sequence method; Test type: Superiority — If the non-inferiority for VRVg-2 versus comparator vaccines was reached at Day 42, then superiority was demonstrated if the overall observed percentage of participants with an RVNA titer >= 0.5 IU/mL at Day 42 was at least 99% in the VRVg-2 Group, with the lower limit of the 95% CI at least 97%; Percentage Difference = 100, 95% CI 2-sided [99.3 to 100]

2. Secondary Outcome: Primary Series: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.5 IU/mL - Pooled Population
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. At Baseline, Group 1 was equivalent to Group 4 (both groups received VRVg-2), Group 2 was equivalent to Group 5 (both groups received Verorab®), and Group 3 was equivalent to Group 6 (both groups received Imovax Rabies®), therefore it was planned to collect and present pooled data of specified Groups, and separately for adults and pediatric participants in this outcome measure.
Time Frame: Cohort 1: Day 0 (pre-vaccination), Day 28 (post-vaccination); Cohort 2: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: Analysis was performed on the PPAS for Day 28. Here, 'overall number of participants analyzed' signifies participants with available data for this outcome measure and 'number analyzed' signifies participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pooled Groups 1 and 4: VRVg-2: Included all pediatric and adult participants of Groups 1 and 4 who received VRVg-2 in Cohort 1 or 2.
- Pooled Groups 2 and 5: Verorab®: Included all pediatric and adult participants of Groups 2 and 5 who received Verorab® in Cohort 1 or 2.
- Pooled Groups 3 and 6: Imovax Rabies®: Included all pediatric and adult participants of Groups 3 and 6 who received Imovax Rabies® in Cohort 1 or 2.
Arm/Group | Pooled Groups 1 and 4: VRVg-2 | Pooled Groups 2 and 5: Verorab® | Pooled Groups 3 and 6: Imovax Rabies®
Number analyzed (Participants) | 861 | 289 | 284
percentage of participants
  Pediatric (< 18 years): number analyzed (Participants) | 266 | 86 | 81
  Pediatric (< 18 years) | 100 [98.6 to 100] | 100 [95.8 to 100] | 100 [95.5 to 100]
  Adult (>= 18 years): number analyzed (Participants) | 595 | 203 | 203
  Adult (>= 18 years) | 98.3 [96.9 to 99.2] | 98.5 [95.7 to 99.7] | 96.6 [93.0 to 98.6]
Statistical Analysis 1: Comparison: Pooled Groups 1 and 4: VRVg-2 vs Pooled Groups 2 and 5: Verorab®; Pooled Groups 1 and 4: VRVg-2 versus Pooled Groups 2 and 5: Verorab®: Pediatric (< 18 years); Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 95% CI of the difference of the percentage between the test groups (Groups 1+4) and control groups (Groups 2+5, Groups 3+6) was > -5% at Day 28; Percentage Difference = 0, 95% CI 2-sided [-1.4 to 4.3]
Statistical Analysis 2: Comparison: Pooled Groups 1 and 4: VRVg-2 vs Pooled Groups 2 and 5: Verorab®; Pooled Groups 1 and 4: VRVg-2 versus Pooled Groups 2 and 5: Verorab®: Adult (>=18 years); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = -0.2, 95% CI 2-sided [-1.9 to 2.7]
Statistical Analysis 3: Comparison: Pooled Groups 1 and 4: VRVg-2 vs Pooled Groups 3 and 6: Imovax Rabies®; Pooled Groups 1 and 4: VRVg-2 versus Pooled Groups 3 and 6: Imovax Rabies®: Pediatric (< 18 years); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 0, 95% CI 2-sided [-1.4 to 4.5]
Statistical Analysis 4: Comparison: Pooled Groups 1 and 4: VRVg-2 vs Pooled Groups 3 and 6: Imovax Rabies®; Pooled Groups 1 and 4: VRVg-2 versus Pooled Groups 3 and 6: Imovax Rabies®: Adult (>= 18 years); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 1.8, 95% CI 2-sided [-0.5 to 5.3]

3. Secondary Outcome: Primary Series: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.5 IU/mL - Pooled Population (Groups 1 and 4) Versus Cohort 1: Group 3: Non-inferiority Analysis
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. At Baseline, Group 1 was equivalent to Group 4 (both groups received VRVg-2), therefore it was planned to collect and present pooled data of specified Group, and separately for adults and pediatric participants in this outcome measure. Data for this outcome measure was planned to be collected at Day 28 for Pooled Groups 1 and 4 and at Day 42 for Primary Series: Cohort-1 Group 3: Imovax Rabies® and reported as overall data for the non-inferiority analysis in this outcome measure.
Time Frame: Pooled Groups 1 and 4: Day 28 (post-vaccination) and Primary Series: Cohort-1 Group 3: Day 42 (post-vaccination)
Population: Analysis was performed on the PPAS that included all participants who received at least 1 dose of the study with no relevant protocol deviation. Here, 'overall number of participants analyzed' signifies participants with available data for this outcome measure and 'number analyzed' signifies participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled Groups 1 and 4: VRVg-2 | Primary Series: Cohort-1 Group 3: Imovax Rabies®
Number analyzed (Participants) | 861 | 162
percentage of participants
  Pediatric (< 18 years): number analyzed (Participants) | 266 | 83
  Pediatric (< 18 years) | 100 [98.6 to 100] | 100 [95.7 to 100]
  Adult (>= 18 years): number analyzed (Participants) | 595 | 79
  Adult (>= 18 years) | 98.3 [96.9 to 99.2] | 100 [95.4 to 100]
Statistical Analysis 1: Comparison: Pooled Groups 1 and 4: VRVg-2 vs Primary Series: Cohort-1 Group 3: Imovax Rabies®; Pooled Groups 1 and 4: VRVg-2 at Day 28 versus Primary Series: Cohort-1 Group 3: Imovax Rabies® at Day 42: Pediatric (< 18 years); Test type: Non-Inferiority — If the non-inferiority objective for VRVg-2 versus comparator vaccines at Day 28 was demonstrated, the overall non-inferiority of 2-dose VRVg-2 at Day 28 versus 3-dose Imovax Rabies® at Day 42 was demonstrated if the non-inferiority between pooled Groups 1+4 and Group 3 were both demonstrated in each age group; Percentage Difference = 0, 95% CI 2-sided [-1.4 to 4.4] — Non-inferiority was demonstrated if the lower limit of the 95% CI of the difference of the percentage between 2-dose VRVg-2 at Day 28 and 3-dose Imovax Rabies® at Day 42 was > -10%
Statistical Analysis 2: Comparison: Pooled Groups 1 and 4: VRVg-2 vs Primary Series: Cohort-1 Group 3: Imovax Rabies®; Pooled Groups 1 and 4: VRVg-2 at Day 28 versus Primary Series: Cohort-1 Group 3: Imovax Rabies® at Day 42: Adult (>= 18 years); Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Percentage Difference = -1.7, 95% CI 2-sided [-3.1 to 3.0] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Primary Series: Groups 1 and 4: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.5 IU/mL - Pooled Population - Superiority Analysis
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. At Baseline, Group 1 was equivalent to Group 4 (both groups received VRVg-2), therefore it was planned to collect and present pooled data of specified Group in this outcome measure.
Time Frame: Day 28 (post-vaccination)
Population: Analysis was performed on the PPAS for Day 28.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled Groups 1 and 4: VRVg-2
Number analyzed (Participants) | 861
percentage of participants | 98.8 [97.9 to 99.4]

5. Secondary Outcome: Primary Series Cohort 1 Group 3: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.5 IU/mL - Non-Inferiority Analysis
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method.
Time Frame: Cohort 1: Day 28 and Day 42 (post-vaccination)
Population: Analysis was performed on the PPAS. Here, 'number analyzed' signifies participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Series: Cohort-1 Group 3: Imovax Rabies®
Number analyzed (Participants) | 162
percentage of participants
  Day 0 | 0 [0 to 2.3]
  Day 28: number analyzed (Participants) | 160
  Day 28 | 98.8 [95.6 to 99.8]
  Day 42 | 100 [97.7 to 100]
Statistical Analysis 1: Comparison: Primary Series: Cohort-1 Group 3: Imovax Rabies®; Imovax Rabies® at Day 28 versus Imovax Rabies® at Day 42; Test type: Non-Inferiority — If the superiority objective of VRVg-2 was reached at Day 28, the non-inferiority of 2-dose Imovax Rabies® at Day 28 versus 3-dose Imovax Rabies® at Day 42 was demonstrated if the lower limit of the 95% CI of the difference of the percentage between the 2-dose Imovax Rabies® at Day 28 and 3-dose Imovax Rabies® at Day 42 was > -10%; Percentage Difference = -1.3, 95% CI 2-sided [-4.4 to 1.3]

6. Secondary Outcome: Primary Series Cohort 1: Rabies Virus Neutralizing Antibody Geometric Mean Titers (GMTs) Against Rabies Virus
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method.
Time Frame: Cohort 1: Day 0 (pre-vaccination), Day 28 and Day 42 (post-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies®
Number analyzed (Participants) | 519 | 169 | 162
IU/mL
  Day 0 | 0.100 [0.100 to 0.100] | 0.101 [0.100 to 0.102] | 0.101 [0.100 to 0.101]
  Day 28: number analyzed (Participants) | 512 | 168 | 160
  Day 28 | 7.16 [6.66 to 7.69] | 4.90 [4.31 to 5.57] | 5.13 [4.48 to 5.87]
  Day 42 | 24.0 [22.4 to 25.7] | 20.0 [17.6 to 22.8] | 16.4 [14.7 to 18.3]

7. Secondary Outcome: Primary Series Cohort 2: Rabies Virus Neutralizing Antibody Geometric Mean Titers (GMTs) Against Rabies Virus
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method.
Time Frame: Cohort 2: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: Analysis was performed on the PPAS for Day 28 that included all participants who received at least 1 dose of the study vaccine in the primary series, with no relevant protocol deviation before Day 28.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies®
Number analyzed (Participants) | 342 | 120 | 124
IU/mL
  Day 0 | 0.101 [0.100 to 0.101] | 0.101 [0.100 to 0.101] | 0.100 [0.100 to 0.101]
  Day 28 | 3.79 [3.42 to 4.20] | 2.92 [2.45 to 3.48] | 3.91 [3.25 to 4.70]

8. Secondary Outcome: Primary Series Cohort 2: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.5 IU/mL
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method.
Time Frame: Cohort 2: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: Analysis was performed on PPAS for Day 28.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies®
Number analyzed (Participants) | 342 | 120 | 124
percentage of participants
  Day 0 | 0 [0.0 to 1.1] | 0 [0.0 to 3.0] | 0 [0.0 to 2.9]
  Day 28 | 97.1 [94.7 to 98.6] | 98.3 [94.1 to 99.8] | 96.0 [90.8 to 98.7]

9. Secondary Outcome: Primary Series Cohort 1: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.2 IU/mL (Lower Limit of Quantification [LLOQ])
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. LLOQ for the RFFIT assay was 0.2 IU/mL.
Time Frame: Cohort 1: Day 0 (pre-vaccination), Day 28 and Day 42 (post-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies®
Number analyzed (Participants) | 519 | 169 | 162
percentage of participants
  Day 0 | 0 [0 to 0.7] | 0 [0 to 2.2] | 0 [0 to 2.3]
  Day 28: number analyzed (Participants) | 519 | 168 | 160
  Day 28 | 100 [99.3 to 100] | 99.4 [96.7 to 100] | 100 [97.7 to 100]
  Day 42 | 100 [99.3 to 100] | 99.4 [96.7 to 100] | 100 [97.7 to 100]

10. Secondary Outcome: Primary Series Cohort 2: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.2 IU/mL (Lower Limit of Quantification [LLOQ])
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. LLOQ for the RFFIT assay was 0.2 IU/mL.
Time Frame: Cohort 2: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: Analysis was performed on the PPAS for Day 28.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies®
Number analyzed (Participants) | 342 | 120 | 124
percentage of participants
  Day 0 | 0 [0 to 1.1] | 0 [0 to 3.0] | 0 [0 to 2.9]
  Day 28 | 99.7 [98.4 to 100] | 100 [97.0 to 100] | 98.4 [94.3 to 99.8]

11. Secondary Outcome: Primary Series Cohort 1: Geometric Mean Titer Ratio (GMTR) of Rabies Virus Neutralizing Antibody Titers
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. GMTRs were calculated as the ratio of GMTs post-vaccination (i.e., on Day 28 and Day 42) and pre-vaccination on Day 0.
Time Frame: Cohort 1: Day 0 (pre-vaccination), Day 28 and Day 42 (post-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies®
Number analyzed (Participants) | 519 | 169 | 162
ratio
  Day 28/Day 0: number analyzed (Participants) | 512 | 168 | 160
  Day 28/Day 0 | 71.5 [66.6 to 76.8] | 48.7 [42.8 to 55.3] | 51.0 [44.6 to 58.3]
  Day 42/Day 0 | 240 [224 to 256] | 199 [174 to 226] | 163 [146 to 182]

12. Secondary Outcome: Primary Series Cohort 2: Geometric Mean Titer Ratio (GMTR) of Rabies Virus Neutralizing Antibody Titers
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. GMTRs were calculated as the ratio of GMTs post-vaccination (i.e., on Day 28) and pre-vaccination on Day 0.
Time Frame: Cohort 2: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: Analysis was performed on the PPAS for Day 28.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies®
Number analyzed (Participants) | 342 | 120 | 124
ratio | 37.7 [34.0 to 41.8] | 29.0 [24.4 to 34.6] | 38.9 [32.4 to 46.7]

13. Secondary Outcome: Primary Series Cohort 1: Percentage of Participants With Determined Complete and Determined Incomplete Virus Neutralization
Description: Virus neutralization was defined as complete (absence of fluorescent cells) and incomplete (presence of fluorescent cells) at the participant/timepoint level at the starting dilution (1/5) of RFFIT assay. Percentage of participants with determined complete and determined incomplete virus neutralization were reported.
Time Frame: Cohort 1: Day 0 (pre-vaccination), Day 28 and Day 42 (post-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies®
Number analyzed (Participants) | 519 | 169 | 162
percentage of participants
  Day 0 - Complete neutralization: number analyzed (Participants) | 504 | 166 | 158
  Day 0 - Complete neutralization | 0.2 [0 to 1.1] | 0.6 [0 to 3.3] | 1.3 [0.2 to 4.5]
  Day 0 - Incomplete neutralization: number analyzed (Participants) | 504 | 166 | 158
  Day 0 - Incomplete neutralization | 99.8 [98.9 to 100] | 99.4 [96.7 to 100] | 98.7 [95.5 to 99.8]
  Day 28 - Complete neutralization: number analyzed (Participants) | 514 | 167 | 161
  Day 28 - Complete neutralization | 100 [99.3 to 100] | 99.4 [96.7 to 100] | 99.4 [96.6 to 100]
  Day 28 - Incomplete neutralization: number analyzed (Participants) | 514 | 167 | 161
  Day 28 - Incomplete neutralization | 0 [0 to 0.7] | 0.6 [0 to 3.3] | 0.6 [0 to 3.4]
  Day 42 - Complete neutralization: number analyzed (Participants) | 518 | 169 | 161
  Day 42 - Complete neutralization | 100 [99.3 to 100] | 99.4 [96.7 to 100] | 100 [97.7 to 100]
  Day 42 - Incomplete neutralization: number analyzed (Participants) | 518 | 169 | 161
  Day 42 - Incomplete neutralization | 0 [0 to 0.7] | 0.6 [0 to 3.3] | 0 [0 to 2.3]

14. Secondary Outcome: Primary Series Cohort 2: Percentage of Participants With Determined Complete and Determined Incomplete Virus Neutralization
Description: as for outcome 13
Time Frame: Cohort 2: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: Analysis was performed on the PPAS for Day 28. Here, 'number analyzed' signifies participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies®
Number analyzed (Participants) | 342 | 120 | 124
percentage of participants
  Day 0 - Complete neutralization: number analyzed (Participants) | 330 | 119 | 117
  Day 0 - Complete neutralization | 0.9 [0.2 to 2.6] | 4.2 [1.4 to 9.5] | 0 [0 to 3.1]
  Day 0 - Incomplete neutralization: number analyzed (Participants) | 330 | 119 | 117
  Day 0 - Incomplete neutralization | 99.1 [97.4 to 99.8] | 95.8 [90.5 to 98.6] | 100 [96.9 to 100]
  Day 28 - Complete neutralization: number analyzed (Participants) | 339 | 120 | 124
  Day 28 - Complete neutralization | 100 [98.9 to 100] | 100 [97.0 to 100] | 98.4 [94.3 to 99.8]
  Day 28 - Incomplete neutralization: number analyzed (Participants) | 339 | 120 | 124
  Day 28 - Incomplete neutralization | 0 [0 to 1.1] | 0 [0 to 3.0] | 1.6 [0.2 to 5.7]

15. Secondary Outcome: Booster Phase: Rabies Virus Neutralizing Antibody (RVNA) Geometric Mean Titers (GMTs) Against Rabies Virus
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. GMTs were expressed in IU/mL.
Time Frame: Month 12 (pre-booster dose) and Month 12 + Day 14 (post-booster dose)
Population: Analysis was performed on PPAS for Booster at Month 12 that included a subset of adults who received a 3 doses regimen and received a single booster dose of VRVg-2 one year after the first vaccination of the primary series (i.e., at Month 12), with no relevant protocol deviation before Month 12 + Day 14.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2): A subset of adult participants who received VRVg-2 vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase at Month 12.
- Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed): A subset of adult participants who received Verorab® vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase at Month 12.
- Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed): A subset of adult participants who received Imovax Rabies® vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase at Month 12.
Arm/Group | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 80 | 26 | 28
IU/mL
  Month 12 | 0.679 [0.526 to 0.878] | 0.540 [0.344 to 0.848] | 0.487 [0.311 to 0.764]
  Month 12 + 14 Days | 56.5 [45.4 to 70.3] | 57.1 [42.6 to 76.7] | 33.7 [22.6 to 50.3]

16. Secondary Outcome: Booster Phase: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.5 IU/mL
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method.
Time Frame: Month 12 (pre-booster dose) and Month 12 + Day 14 (post-booster dose)
Population: Analysis was performed on the PPAS for Booster at Month 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 80 | 26 | 28
percentage of participants
  Month 12 | 53.8 [42.2 to 65.0] | 53.8 [33.4 to 73.4] | 35.7 [18.6 to 55.9]
  Month 12 + 14 days | 100 [95.5 to 100] | 100 [86.8 to 100] | 100 [87.7 to 100]

17. Secondary Outcome: Booster Phase: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.2 IU/mL (LLOQ)
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. LLOQ for the RFFIT assay was 0.2 IU/mL.
Time Frame: Month 12 (pre-booster dose) and Month 12 + Day 14 (post-booster dose)
Population: Analysis was performed on the PPAS for Booster at Month 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 80 | 26 | 28
percentage of participants
  Month 12 | 86.3 [76.7 to 92.9] | 76.9 [56.4 to 91.0] | 85.7 [67.3 to 96.0]
  Month 12 + 14 days | 100 [95.5 to 100] | 100 [86.8 to 100] | 100 [87.7 to 100]

18. Secondary Outcome: Booster Phase: Geometric Mean Titer Ratio (GMTR) of Rabies Virus Neutralizing Antibody Titers
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. GMTRs were calculated as the ratio of GMTs post vaccination (i.e., on Month 12 and Month 12 + Day 14) and pre-vaccination on Day 0, pre-booster dose on Month 12.
Time Frame: Day 0 (pre-vaccination), Month 12 (pre-booster dose) and Month 12 + Day 14 (post-booster dose)
Population: Analysis was performed on the PPAS for Booster at Month 12.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 80 | 26 | 28
ratio
  Month 12/Day 0 | 6.79 [5.26 to 8.78] | 5.40 [3.44 to 8.48] | 4.78 [3.10 to 7.37]
  Month 12+14 days/Day 0 | 565 [454 to 703] | 571 [426 to 767] | 331 [219 to 500]
  Month 12+14 days/Month 12 | 83.2 [62.0 to 112] | 106 [62.7 to 178] | 69.2 [39.6 to 121]

19. Secondary Outcome: Booster Phase: Percentage of Participants With Determined Complete and Determined Incomplete Virus Neutralization
Description: as for outcome 13
Time Frame: Month 12 (pre-booster dose) and Month 12 + Day 14 (post-booster dose)
Population: Analysis was performed on the PPAS for Booster at Month 12. Here, 'number analyzed' signifies participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 80 | 26 | 28
percentage of participants
  Month 12 - Complete neutralization: number analyzed (Participants) | 77 | 25 | 23
  Month 12 - Complete neutralization | 96.1 [89.0 to 99.2] | 84.0 [63.9 to 95.5] | 95.7 [78.1 to 99.9]
  Month 12 - Incomplete neutralization: number analyzed (Participants) | 77 | 25 | 23
  Month 12 - Incomplete neutralization | 3.9 [0.8 to 11.0] | 16.0 [4.5 to 36.1] | 4.3 [0.1 to 21.9]
  Month 12 + 14 days - Complete neutralization: number analyzed (Participants) | 80 | 26 | 27
  Month 12 + 14 days - Complete neutralization | 100 [95.5 to 100] | 100 [86.8 to 100] | 100 [87.2 to 100]
  Month 12 + 14 days - Incomplete neutralization: number analyzed (Participants) | 80 | 26 | 27
  Month 12 + 14 days - Incomplete neutralization | 0 [0 to 4.5] | 0 [0 to 13.2] | 0 [0 to 12.8]

20. Secondary Outcome: Booster Phase Cohort 2: Rabies Virus Neutralizing Antibody (RVNA) Geometric Mean Titers (GMTs) Against Rabies Virus
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. GMTs were expressed in International units/milliliter (IU/mL).
Time Frame: Month 24 up to Month 36 (pre-booster dose) and Month 24 up to Month 36 + Day 14 (post-booster dose)
Population: Results are based on the PPAS for booster between Month 24 up to Month 36 that included a subset of adults who received a 1 week 2-dose regimen and a single booster dose of VRVg-2 between Month 24 and up to Month 36 after the first vaccination of the primary series with no relevant protocol deviation before Month 24 up to Month 36 + Day 14.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2): A subset of adult participants who received VRVg-2 vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase between Month 24 up to Month 36.
- Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed): A subset of adult participants who received Verorab® vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase between Month 24 up to Month 36.
- Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed): A subset of adult participants who received Imovax Rabies® vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase between Month 24 up to Month 36.
Arm/Group | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 108 | 33 | 37
IU/mL
  Month 24 up to Month 36 | 0.761 [0.607 to 0.953] | 0.536 [0.385 to 0.747] | 0.903 [0.603 to 1.35]
  Month 24 up to Month 36 + 14 Days | 95.4 [76.7 to 119] | 89.4 [55.8 to 143] | 64.7 [43.7 to 95.9]

21. Secondary Outcome: Booster Phase Cohort 2: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.5 IU/mL
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. Percentages are rounded off to the tenth decimal place.
Time Frame: Month 24 up to Month 36 (pre-booster dose) and Month 24 up to Month 36 + Day 14 (post-booster dose)
Population: Results are based on the PPAS for booster between Month 24 up to Month 36.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 108 | 33 | 37
percentage of participants
  Month 24 up to Month 36 | 62.0 [52.2 to 71.2] | 51.5 [33.5 to 69.2] | 64.9 [47.5 to 79.8]
  Month 24 up to Month 36 + 14 Days | 100 [96.6 to 100] | 100 [89.4 to 100] | 100 [90.5 to 100]

22. Secondary Outcome: Booster Phase Cohort 2: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.2 IU/mL (Lower Limit of Quantification [LLOQ])
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. LLOQ for the RFFIT assay was 0.2 IU/mL. Percentages are rounded off to the tenth decimal place.
Time Frame: Month 24 up to Month 36 (pre-booster dose) and Month 24 up to Month 36 + Day 14 (post-booster dose)
Population: Results are based on the PPAS for booster between Month 24 up to Month 36.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 108 | 33 | 37
percentage of participants
  Month 24 up to Month 36 | 89.8 [82.5 to 94.8] | 87.9 [71.8 to 96.6] | 89.2 [74.6 to 97.0]
  Month 24 up to Month 36 + 14 Days | 100 [96.6 to 100] | 100 [89.4 to 100] | 100 [90.5 to 100]

23. Secondary Outcome: Booster Phase Cohort 2: Geometric Mean Titer Ratio (GMTR) of Rabies Virus Neutralizing Antibody Titers
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. GMTRs were calculated as the ratio of GMTs pre-booster/pre-vaccination (Month 24 up to Month 36/Day 0); post-booster/pre-vaccination (Month 24 up to Month 36 +14 days/Day 0); post-booster/pre-booster (Month 24 up to Month 36+14 days/Month 24 up to Month 36).
Time Frame: Day 0 (pre-vaccination), Month 24 up to Month 36 (pre-booster dose) and Month 24 up to Month 36 + Day 14 (post-booster dose)
Population: Results are based on the PPAS for booster between Month 24 up to Month 36.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 108 | 33 | 37
ratio
  Month 24 up to Month 36/Day 0 | 7.58 [6.06 to 9.48] | 5.30 [3.80 to 7.40] | 9.03 [6.03 to 13.5]
  Month 24 up to Month 36 +14 days/Day 0 | 951 [764 to 1184] | 885 [548 to 1430] | 647 [437 to 959]
  Month 24 up to Month 36+14 days/Month 24 up to Month 36 | 125 [98.1 to 160] | 167 [101 to 276] | 71.7 [42.3 to 122]

24. Secondary Outcome: Booster Phase Cohort 2: Percentage of Participants With Determined Complete and Determined Incomplete Virus Neutralization
Description: Virus neutralization was defined as complete (absence of fluorescent cells) and incomplete (presence of fluorescent cells) at the participant/timepoint level at the starting dilution (1/5) of RFFIT assay. Percentage of participants with determined complete and determined incomplete virus neutralization were reported. Percentages are rounded off to the tenth decimal place.
Time Frame: Month 24 up to Month 36 (pre-booster dose) and Month 24 up to Month 36 + Day 14 (post-booster dose)
Population: Results are based on the PPAS for Booster between Month 24 up to Month 36. Here, 'number analyzed' signifies number of participants with available data for this outcome measure for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 108 | 33 | 37
percentage of participants
  Month 24 up to Month 36- Complete neutralization: number analyzed (Participants) | 107 | 33 | 37
  Month 24 up to Month 36- Complete neutralization | 94.1 [87.5 to 97.8] | 93.8 [79.2 to 99.2] | 91.9 [78.1 to 98.3]
  Month 24 up to Month 36- Incomplete neutralization: number analyzed (Participants) | 107 | 33 | 37
  Month 24 up to Month 36- Incomplete neutralization | 5.9 [2.2 to 12.5] | 6.3 [0.8 to 20.8] | 8.1 [1.7 to 21.9]
  Month 24 up to Month 36 + 14 days- Complete neutralization | 100 [96.6 to 100] | 100 [89.4 to 100] | 100 [90.5 to 100]
  Month 24 up to Month 36 + 14 days- Incomplete neutralization | 0 [0 to 3.4] | 0 [0 to 10.6] | 0 [0 to 9.5]

25. Secondary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study vaccine and does not necessarily had to have a causal relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset post-vaccination. All participants were observed for 30 minutes after any vaccination, and any unsolicited AEs occurred during that time were recorded as immediate unsolicited AEs in the CRB.
Time Frame: Within 30 minutes after any vaccination
Population: Analysis was performed on the safety analysis set (SafAS) that included participant who had received at least one dose of the study vaccine and were analyzed according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Series: Cohort-1 Group 1: VRVg-2: Pediatric and adult participants received 3 intramuscular (IM) injections of VRVg-2 vaccine at Day 0, Day 7, and Day 28 respectively.
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies® | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies® | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 607 | 202 | 200 | 419 | 139 | 139 | 94 | 31 | 32
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Booster Phase Cohort 2: Number of Participants With Immediate Unsolicited Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study vaccine and does not necessarily had to have a causal relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRB in terms of diagnosis and/or onset post-vaccination. All participants were observed for 30 minutes after any vaccination, and any unsolicited AEs occurred during that time were recorded as immediate unsolicited AEs in the CRB.
Time Frame: Within 30 minutes after any vaccination
Population: Results are based on the SafAS that included participants who had received at least one dose of the study vaccine and were analyzed according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 128 | 41 | 43
Participants | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Systemic Reactions
Description: A SR was an expected AR observed and reported under conditions (nature and onset) pre-listed (i.e., solicited) in the protocol and CRB and considered as related to vaccination. An AR was all noxious and unintended responses to a medicinal product related to any dose. Solicited systemic reactions included fever, vomiting, crying abnormal, drowsiness, appetite loss, irritability, headache, malaise and myalgia. Solicited systemic reactions were collected by different age groups: Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability were collected for participants aged 12 to 23 months. Fever, Headache, Malaise and Myalgia were collected for participants aged >= 2 years.
Time Frame: Within 7 Days after any vaccination
Population: Analysis was performed on the SafAS. Here, 'number analyzed' signifies participants with available data for each specified category and "0" in the number analyzed denotes that data was not collected and analyzed for the specified category as no pediatric participants were available for analysis in the specified groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies® | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies® | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 607 | 202 | 200 | 419 | 139 | 139 | 94 | 31 | 32
Participants
  Fever: number analyzed (Participants) | 606 | 201 | 200 | 419 | 139 | 139 | 94 | 31 | 32
  Fever | 50 | 11 | 4 | 2 | 0 | 0 | 0 | 0 | 0
  Vomiting: number analyzed (Participants) | 17 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting | 4 | 1 | 1 |  |  |  |  |  |
  Crying abnormal: number analyzed (Participants) | 17 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Crying abnormal | 8 | 0 | 1 |  |  |  |  |  |
  Drowsiness: number analyzed (Participants) | 17 | 202 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Drowsiness | 4 | 1 | 0 |  |  |  |  |  |
  Appetite lost: number analyzed (Participants) | 17 | 202 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Appetite lost | 3 | 1 | 0 |  |  |  |  |  |
  Irritability: number analyzed (Participants) | 17 | 202 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Irritability | 8 | 1 | 0 |  |  |  |  |  |
  Headache: number analyzed (Participants) | 590 | 199 | 198 | 419 | 139 | 139 | 94 | 31 | 32
  Headache | 128 | 49 | 46 | 39 | 9 | 8 | 4 | 3 | 5
  Malaise: number analyzed (Participants) | 590 | 199 | 198 | 419 | 139 | 139 | 94 | 31 | 32
  Malaise | 161 | 45 | 48 | 37 | 10 | 12 | 8 | 3 | 7
  Myalgia: number analyzed (Participants) | 590 | 199 | 198 | 419 | 139 | 139 | 94 | 31 | 32
  Myalgia | 249 | 66 | 78 | 78 | 12 | 29 | 23 | 9 | 15

28. Secondary Outcome: Booster Phase Cohort 2: Number of Participants With Systemic Reactions
Description: as for outcome 27
Time Frame: Within 7 Days after any vaccination
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 128 | 41 | 43
Participants
  Fever | 0 | 0 | 0
  Vomiting: number analyzed (Participants) | 0 | 0 | 0
  Crying abnormal: number analyzed (Participants) | 0 | 0 | 0
  Drowsiness: number analyzed (Participants) | 0 | 0 | 0
  Appetite lost: number analyzed (Participants) | 0 | 0 | 0
  Irritability: number analyzed (Participants) | 0 | 0 | 0
  Headache | 3 | 0 | 0
  Malaise | 5 | 1 | 0
  Myalgia | 10 | 0 | 0

29. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: A solicited reaction (SR) was an expected AR observed and reported under conditions (nature and onset) pre-listed (i.e., solicited) in the protocol and CRB and considered as related to vaccination. An AR was all noxious and unintended responses to a medicinal product related to any dose. Solicited injection site reactions included tenderness/pain, erythema and swelling.
Time Frame: Within 7 Days after any vaccination
Population: Analysis was performed on the SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies® | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies® | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 607 | 202 | 200 | 419 | 139 | 139 | 94 | 31 | 32
Participants
  Injection site tenderness/pain | 344 | 95 | 106 | 111 | 30 | 43 | 44 | 12 | 17
  Injection site erythema | 24 | 6 | 6 | 0 | 0 | 1 | 0 | 0 | 0
  Injection site swelling | 14 | 4 | 13 | 1 | 0 | 1 | 0 | 1 | 0

30. Secondary Outcome: Booster Phase Cohort 2: Number of Participants With Solicited Injection Site Reactions
Description: A SR was an expected AR observed and reported under conditions (nature and onset) pre-listed (i.e., solicited) in the protocol and CRB and considered as related to vaccination. An AR was all noxious and unintended responses to a medicinal product related to any dose. Solicited injection site reactions included tenderness/pain, erythema and swelling.
Time Frame: Within 7 Days after any vaccination
Population: Results are based on the SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 128 | 41 | 43
Participants
  Injection site tenderness/pain | 20 | 2 | 6
  Injection site erythema | 0 | 0 | 0
  Injection site swelling | 0 | 0 | 0

31. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An AE was defined as any untoward medical occurrence in a participant who received study vaccine and does not necessarily had to have a causal relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions pre-listed in the CRB in terms of diagnosis and/or onset post-vaccination.
Time Frame: Within 28 Days after any vaccination
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies® | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies® | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 607 | 202 | 200 | 419 | 139 | 139 | 94 | 31 | 32
Participants | 137 | 45 | 40 | 44 | 18 | 12 | 13 | 3 | 5

32. Secondary Outcome: Booster Phase Cohort 2: Number of Participants With Unsolicited Adverse Events
Description: as for outcome 31
Time Frame: Within 28 Days after any vaccination
Population: Results are based on the SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 128 | 41 | 43
Participants | 15 | 1 | 3

33. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: An SAEs was any untoward medical occurrence that at any dose resulted in death, life-threatening, initial or prolonged inpatient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect or a medically important event. An AESI was defined as one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor was appropriate. All SAEs and AESIs occurring during the study that were related to the product administered were reported by the Investigator to the Independent Ethics Committee/Institutional Review Board. Relatedness to study vaccine was based on Investigator's discretion.
Time Frame: From Baseline (Day 0) up to 6 months after last vaccination (i.e., up to 7 months for Primary Series Cohorts 1 & 2 and up to Month 18 for Booster Phase, Cohort 1)
Population: Analysis was performed on SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies® | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies® | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 607 | 202 | 20 | 419 | 139 | 139 | 94 | 31 | 32
Participants
  SAEs | 10 | 3 | 5 | 2 | 0 | 1 | 2 | 0 | 1
  AESIs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

34. Secondary Outcome: Booster Phase Cohort 2: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: as for outcome 33
Time Frame: From Baseline (Day 0) up to 6 months after last vaccination (i.e., up to Month 42)
Population: Results are based on the SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed)
Number analyzed (Participants) | 128 | 41 | 43
Participants
  SAEs | 3 | 0 | 1
  AESIs | 0 | 0 | 0

35. Primary Outcome: Primary Series Cohort 1: Percentage of Participants With Rabies Virus Neutralizing Antibody (RVNA) Titer Greater Than or Equal to (>=) 0.5 IU/mL
Description: RVNA titer against rabies virus was assessed using the Rapid Fluorescent Focus Inhibition test (RFFIT) assay method.
Time Frame: Day 42 (post-vaccination)
Population: Analysis was performed on the per-protocol analysis set (PPAS) for Day 42 that included all participants who received at least 1 dose of the study vaccine in the primary series, with no relevant protocol deviation before Day 42. Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was planned to be collected and analyzed only for Primary series cohort-1 and separately for adults and pediatric participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies®
Number analyzed (Participants) | 519 | 169 | 162
percentage of participants
  Pediatric (< 18 years): number analyzed (Participants) | 265 | 85 | 83
  Pediatric (< 18 years) | 100 [98.6 to 100] | 100 [95.8 to 100] | 100 [95.7 to 100]
  Adult (>= 18 years): number analyzed (Participants) | 254 | 84 | 79
  Adult (>= 18 years) | 100 [98.6 to 100] | 98.8 [93.5 to 100] | 100 [95.4 to 100]
Statistical Analysis 1: Comparison: Primary Series: Cohort-1 Group 1: VRVg-2 vs Primary Series: Cohort-1 Group 2: Verorab®; Primary Series: Cohort-I Group 1: VRVg-2 versus Primary Series: Cohort-I Group 2: Verorab®: Pediatric (< 18 years); Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 95 percent (%) confidence interval (CI) of the difference of the percentages between the test group (Group 1) and control groups (Group 2, Group 3) was greater than (>) -5% at Day 42; Percentage Difference = 0, 95% CI 2-sided [-1.4 to 4.3]
Statistical Analysis 2: Comparison: Primary Series: Cohort-1 Group 1: VRVg-2 vs Primary Series: Cohort-1 Group 2: Verorab®; Primary Series: Cohort-I Group 1: VRVg-2 versus Primary Series: Cohort-I Group 2: Verorab®: Adult (>=18 years); Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 95% CI of the difference of the percentages between the test group (Group 1) and control groups (Group 2, Group 3) was > -5% at Day 42; Percentage Difference = 1.2, 95% CI 2-sided [-0.6 to 6.4]
Statistical Analysis 3: Comparison: Primary Series: Cohort-1 Group 1: VRVg-2 vs Primary Series: Cohort-1 Group 3: Imovax Rabies®; Primary Series: Cohort-I Group 1: VRVg-2 versus Primary Series: Cohort-I Group 3: Imovax Rabies: Pediatric (< 18 years); Test type: Non-Inferiority — [test comment as in outcome 35, analysis 2]; Percentage Difference = 0, 95% CI 2-sided [-1.4 to 4.4]
Statistical Analysis 4: Comparison: Primary Series: Cohort-1 Group 1: VRVg-2 vs Primary Series: Cohort-1 Group 3: Imovax Rabies®; Primary Series: Cohort-I Group 1: VRVg-2 versus Primary Series: Cohort-I Group 3: Imovax Rabies: Adult (>= 18 years); Test type: Non-Inferiority — [test comment as in outcome 35, analysis 2]; Percentage Difference = 0, 95% CI 2-sided [-1.5 to 4.6]

ADVERSE EVENTS:
Time Frame: From Baseline (Day 0) up to 6 months after last vaccination (i.e., up to 7 months for Primary Series Cohorts 1 and 2 and up to Month 18 for Booster Phase Cohort 1, and up to Month 42 for Booster Phase Cohort 2).
Description: SafAS. SR: expected AR observed and reported under conditions (nature and onset) pre-listed (i.e., solicited) in protocol and CRB. Unsolicited AE: observed AE that did not fulfill conditions pre-listed (i.e., solicited) in the CRB in terms of diagnosis and/or onset post-vaccination. In the AE section, SR fever is reported as pyrexia. AE data is based on the SafAS.
Groups:
- Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2): A subset of adult participants who received 3 IM injections of VRVg-2 vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase at Month 12.
- Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed): A subset of adult participants who received 3 IM injections of Verorab® vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase at Month 12.
- Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed): A subset of adult participants who received 3 IM injections of Imovax Rabies® vaccination in primary series and completed the follow-up period received a booster injection of VRVg-2 in the booster phase at Month 12.
- Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2): A subset of adult participants who received VRVg-2 vaccination in primary series and completed the follow-up period received a booster injection ofVRVg-2 in the booster phase between Month 24 up to Month 36.
Arm/Group | Primary Series: Cohort-1 Group 1: VRVg-2 | Primary Series: Cohort-1 Group 2: Verorab® | Primary Series: Cohort-1 Group 3: Imovax Rabies® | Primary Series: Cohort-2 Group 4: VRVg-2 | Primary Series: Cohort-2 Group 5: Verorab® | Primary Series: Cohort-2 Group 6: Imovax Rabies® | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed) | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed)
All-Cause Mortality (participants affected / at risk) | 0/607 | 0/202 | 0/200 | 0/419 | 0/139 | 0/139 | 0/94 | 0/31 | 0/32 | 0/128 | 0/41 | 0/43
Serious Adverse Events (participants affected / at risk) | 10/607 | 3/202 | 5/200 | 2/419 | 0/139 | 1/139 | 2/94 | 0/31 | 1/32 | 3/128 | 0/41 | 1/43
Other Adverse Events (participants affected / at risk) | 414/607 | 121/202 | 128/200 | 130/419 | 34/139 | 48/139 | 48/94 | 15/31 | 18/32 | 21/128 | 2/41 | 6/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Series: Cohort-1 Group 1: VRVg-2 (N=607) | Primary Series: Cohort-1 Group 2: Verorab® (N=202) | Primary Series: Cohort-1 Group 3: Imovax Rabies® (N=200) | Primary Series: Cohort-2 Group 4: VRVg-2 (N=419) | Primary Series: Cohort-2 Group 5: Verorab® (N=139) | Primary Series: Cohort-2 Group 6: Imovax Rabies® (N=139) | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) (N=94) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) (N=31) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed) (N=32) | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) (N=128) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) (N=41) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed) (N=43)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup Infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue Fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious Mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exposure To Communicable Disease (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratorhexis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma Of The Cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Imminent Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Series: Cohort-1 Group 1: VRVg-2 (N=607) | Primary Series: Cohort-1 Group 2: Verorab® (N=202) | Primary Series: Cohort-1 Group 3: Imovax Rabies® (N=200) | Primary Series: Cohort-2 Group 4: VRVg-2 (N=419) | Primary Series: Cohort-2 Group 5: Verorab® (N=139) | Primary Series: Cohort-2 Group 6: Imovax Rabies® (N=139) | Booster Phase: Cohort-1 Group 1: VRVg-2 (Primed With VRVg-2) (N=94) | Booster Phase: Cohort-1 Group 2: VRVg-2 (Verorab® Primed) (N=31) | Booster Phase: Cohort-1 Group 3: VRVg-2 (Imovax Rabies® Primed) (N=32) | Booster Phase: Cohort-2 Group 4: VRVg-2 (Primed With VRVg-2) (N=128) | Booster Phase: Cohort-2 Group 5: VRVg-2 (Verorab® Primed) (N=41) | Booster Phase:Cohort-2 Group 6: VRVg-2 (Imovax Rabies® Primed) (N=43)
Injection Site Pain (General disorders) | 344 (655) | 95 (158) | 106 (191) | 111 (167) | 30 (41) | 43 (63) | 44 (44) | 12 (12) | 17 (17) | 20 (20) | 2 (2) | 6 (6)
Injection Site Swelling (General disorders) | 14 (19) | 4 (4) | 13 (18) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 161 (229) | 45 (57) | 48 (79) | 37 (43) | 10 (14) | 12 (16) | 8 (8) | 3 (3) | 7 (7) | 5 (5) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 51 (54) | 12 (12) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 27 (27) | 9 (9) | 12 (14) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 249 (405) | 67 (103) | 79 (135) | 78 (103) | 12 (17) | 30 (38) | 24 (24) | 9 (9) | 15 (15) | 10 (10) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 130 (178) | 50 (66) | 47 (62) | 40 (46) | 10 (14) | 8 (9) | 4 (4) | 3 (3) | 7 (7) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT04127786/Prot_002.pdf
  • Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT04127786/SAP_003.pdf